CLINICAL TRIAL: NCT04120844
Title: Effectiveness of Motivational Interviewing on Improving Care for Patients With Type 2 Diabetes in China: A Randomized Controlled Trial
Brief Title: Effectiveness of Motivational Interviewing on Improving Care for Type 2 Diabetes Mellitus Patients in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JCYJ20150331142757385
Record Dates: First submitted 2019-09-26; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Diabete Type 2
Keywords: Type 2 diabete; Motivational interviewing; Patient empowerment; Self-management; China
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Participation | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group (n=117) received a four-session PEP in small groups over one month by trained nurses and doctors.
  Interventions: Behavioral: Motivational interviewing (MI)-based patient empowerment program (PEP)
- Control (Placebo Comparator): The control group (n=108) received the traditional lecture-style health education on Diabetes Mellitus.
  Interventions: Behavioral: Traditional lecture style health education

INTERVENTIONS:
Behavioral: Motivational interviewing (MI)-based patient empowerment program (PEP) — Motivational interviewing (MI) is a collaborative, patient-centered counseling approach that aims to elicit behavior change. Counselors use empathy and other techniques to create an atmosphere to help patients to explore the discrepancies between the goals and their current behavior. The focus of MI is to find and resolve the ambivalence, improve patients' perception of the importance of behavior change, and support them to make the change. MI provides a structural framework with guiding principles that can be easily followed by the primary care doctors. Program content was further informed by the Hospital Authority Patient Empowerment Program in Hong Kong. The education program consisted of four modules, held once a week, that each lasted approximately 1½ to 2 hours. They were grouped under the following four broad headings: Knowing Diabetes, Diabetes Self-Care, Healthy Diet and Physical Exercise.
  Arms: Intervention
Behavioral: Traditional lecture style health education — The control group received traditional lectures that consisted solely of conveying healthcare information to patients. In order to minimize intervention bias, the control group lectures were standardized and adapted into four modules, namely knowing diabetes, healthy diet, physical exercises, and how to use medication correctly, which were similar topic headings, durations and frequencies to those of the intervention group. Each lecture was 1 hour and was provided by one of four health professionals (a pharmacist, dietician, endocrinologist or nurse) who had never received any prior training in MI. We consciously avoided the inclusion of elements of self-reflection and motivation in these lectures.
  Arms: Control

SUMMARY:
The International Diabetes Federation estimated that there were nearly 110 million diabetes mellitus (DM) patients in China, which was the highest number recorded in the world. In response to the rising patient numbers and costs, the Chinese government has invested heavily in primary healthcare, with the goal of improving chronic disease management in the primary care settings. A key part of the primary care improvement program prioritizes health education as a route to lifestyle modification. Although the content and modes of delivery vary enormously, most of the programs focused on providing information rather than facilitating patient change. The impacts of traditional patient education on lifestyle modification and changes in psychological status have been reported to be suboptimal. It is therefore necessary to rethink and explore a more structured, patient-centered approach to health education at improving the outcomes of DM control.

Motivational interviewing (MI) is a collaborative, patient-centered counseling approach that aims to elicit behavior change.The focus of MI is to find and resolve the ambivalence, improve patients' perception of the importance of behavior change, and support them to make the change. MI provides a structural framework with guiding principles that can be easily followed by the primary care doctors. Some studies show that MI can contribute to improve healthy eating, weight control and increases in physical activity, but most research focused on intermediate outcome measures and did not evaluate the readiness to change. MI can be utilized by a variety of healthcare providers, which makes it adaptable for different culture and clinical settings. The effectiveness of MI in Chinese diabetic patients remains uncertain.Therefore, in this study, we adopted the group MI approach and developed a patient empowerment program (PEP) utilizing the techniques and framework of MI. We compared this to the most common form of DM education in China, a lecture on DM to patients and their carers in a hospital lecture theatre in a didactic manner. The study aimed to assess the effectiveness of the MI approach in terms of patient lifestyle modification and improving DM controls compared to the control group in a non-blinded randomized controlled trial (RCT) design.

DETAILED DESCRIPTION:
This RCT was implemented from May 2016 to April 2017 in Shenzhen, China. Shenzhen is the fourth-biggest city in China, with a rapidly expanding population of 12 million people and the highest GDP in the country. Most DM patients in China are managed at Endocrine Specialist hospital clinics, while the more stable patients are treated in the community. Therefore, we chose an endocrine specialist outpatient clinic and a family medicine clinic at the University of Hong Kong-Shenzhen Hospital (HKU-SZH), as well as three community health centers in the Luohu district as the sampling frame. DM patients were recruited by doctors at consultations. This is because health education lectures are one of the routine diabetes management strategies used by healthcare providers in China and patients are normally invited by their doctors to attend these lectures.

Sample size estimation was calculated based on the previous published research conducted elsewhere in which the DM patients were given MI-guided behavior change counselling. The "Problem Areas in Diabetes" (PAID) score in that study was 29±22.64 in the intervention group vs. 29±24.32 in the control group. Therefore, 192 participants were needed to detect 10% effect size with an alpha of 0.05 and a power of 80.0%. With 15% of loss to follow-up anticipated, a total of 225 participants were targeted.

Descriptive statistics were used to summarize characteristics of the participants. We analyzed the baseline data of the intervention and control groups to determine the consistency of the characteristics across the two groups of patients. The t-test was used for continuous variables such as waist circumference, body weight, and BMI, whereas chi-squared test was used for categorical variables in stages of change such as smoking, drinking, and exercise. Changes in PAID and PEI in post-intervention and follow-ups between the two groups were calculated and tested.

When analyzing the two sets of variables in the intervention and control groups, we followed the principle of intent-to-treat analysis i.e. if the participant failed to participate in all four modules, the first questionnaire results would be assumed and analyzed as the final data, using the mixed design analysis of variance. In detecting the relationship between the continuity variable and categorical variable, we used bivariate correlation analyses. All analyses were performed in SPSS 20.0. We used p value<0.05 as the cut-off point of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c between 7-10%
* 18-75 years old
* No known severe comorbidities or complications, such as cancer, unstable angina, frequent exacerbation of chronic obstructive pulmonary disease, or diabetic retinopathy
* Cognitively competent enough to understand written and the oral expression of the language native to the study site

Exclusion Criteria:

* Known severe comorbidities or complications, such as cancer, unstable angina, frequent exacerbation of chronic obstructive pulmonary disease, or diabetic retinopathy
* Illiterate, or cognitively competent enough to understand written and the oral expression of the language native to the study site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Problem Areas in Diabetic (PAID) Questionnaire | 3 months
  PAID is a self-administered 20-item scale. Each item is scored from 0 (not a problem) to 4 (serious problem). The sum of all item scores multiplied by 1.25 gives the total PAID score, which ranges from 0 to 100, higher scores reflecting greater emotional distress. A score of 40 or above is indicative of severe emotional distress.

SECONDARY OUTCOMES:
"Patient Enablement Index" (PEI) score | 3 months
  The PEI is a scale that measures patients' enablement, it was also used to measure patient enablement in this study.Subjects with PEI total score> 0 are considered to have enablement over the past 12-month period, while those with PEI total score = 0 were considered to have no enablement over the period. The PEI scale had been validated in the Chinese population.
Stages of Change score | 3 months
  Motivation for lifestyle change was measured in this study based on the "Stages of Change" model to assess participants' readiness to change in behaviors such as smoking, drinking or exercise and their adherence to treatment. The mean stage-of-change score may be a more stable estimate of stage of change.

CONTACTS AND LOCATIONS:
Overall Officials: Jingya Yan, Principal Investigator — The University of Hong Kong-Shenzhen Hospital; Wei Liang, Principal Investigator — The University of Hong Kong - Shenzhen Hospital, Shenzhen, China.; Chen Qingqi, Principal Investigator — The University of Hong Kong-Shenzhen Hospital; Wong Chi Wai William, Principal Investigator — The University of Hong Kong-Shenzhen Hospital; Jennifer Li, Principal Investigator — The University of Hong Kong-Shenzhen Hospital

IPD SHARING:
Plan to Share IPD: Yes
Subject to principal investigator's approval
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Li Z, Chen Q, Yan J, Liang W, Wong WCW. Effectiveness of motivational interviewing on improving Care for Patients with type 2 diabetes in China: A randomized controlled trial. BMC Health Serv Res. 2020 Jan 23;20(1):57. doi: 10.1186/s12913-019-4776-8. PMID 31973759